CLINICAL TRIAL: NCT01772355
Title: Effectiveness and Possible Complications of Core Needle Biopsy of Orbital Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yarovoy Andrey (Other Government)
Responsible Party: Sponsor-Investigator, Yarovoy Andrey, MD, PhD, head ocular oncology department, The S.N. Fyodorov Eye Microsurgery State Institution
Organization: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: core biopsy of orbital tumors
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Orbial Mass Lesion
Keywords: orbit; tumor; core biopsy
MeSH Terms: conditions — Neoplasms

ARMS (1):
- tissue core (Other): semi automated core needle biopsy of the orbital tumors
  Interventions: Device: semi automated core needle biopsy of orbital tumors

INTERVENTIONS:
Device: semi automated core needle biopsy of orbital tumors

SUMMARY:
Core needle biopsy of orbital mass lesions with a semiautomated needles is a safe procedure that provides a sufficient amount of tissue material for standard histological and immunohistochemical analysis and can be an alternative or supplement to fine needle aspiration biopsy

ELIGIBILITY:
Inclusion Criteria:

* unresectable mass lesions with diffuse involvement of the orbit or the tumors with infiltrative growth and indistinct borders which needed to have morphologic verification

Exclusion Criteria:

* An anti-coagulant therapy at the time of biopsy,
* bleeding diathesis,
* suspected hypervascular lesions,
* orbital roof destruction with a tumor,
* apical location of the tumor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
true identification of an orbital tumor with a core needle biopsy | five years

CONTACTS AND LOCATIONS:
Locations (1):
- The S.Fyodorov Eye Microsurgery Federal State Institution, Moscow, Russia

REFERENCES:
- [Derived] Yarovoy AA, Bulgakova ES, Shatskikh AV, Uzunyan DG, Kleyankina SS, Golubeva OV. CORE needle biopsy of orbital tumors. Graefes Arch Clin Exp Ophthalmol. 2013 Aug;251(8):2057-61. doi: 10.1007/s00417-013-2315-6. Epub 2013 Mar 21. PMID 23515750